CLINICAL TRIAL: NCT05700812
Title: Feasibility Study of IUD Placement Without Sounding
Brief Title: IUD Placement Without Sounding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1952890
Record Dates: First submitted 2022-12-22; First posted 2023-01-26 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2023-06

CONDITIONS: IUD; IUD Insertion Complication; IUD; Complications

STUDY DESIGN:
Intervention Model Description: Three phase study. Phase one will only include gathering baseline data without intervention. Phases two and three each include a different intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IUD insertion study in three phases (Experimental): In phase one, the IUD will be placed in standard fashion with a uterine sound to obtain baseline data.
  In phase two, the IUD will be placed without the use of a uterine sound and under abdominal ultrasound guidance.
  In phase three, the IUD will be placed without the use of a uterine sound and without ultrasound guidance.
  Interventions: Procedure: Sound sparing levonorgestrel 52 mg IUD placement

INTERVENTIONS:
Procedure: Sound sparing levonorgestrel 52 mg IUD placement — In phase one, the IUD will be placed in a standard fashion with the use of a uterine sound to obtain baseline data.
  In the experimental phases of the study (phase 2 and 3) the levonorgestrel 52 mg IUD will be placed without the use of a uterine sound. In phase 2 the IUD will be placed under abdominal ultrasound guidance. In phase 3 the IUD will be placed without abdominal ultrasound guidance.

SUMMARY:
The purpose of this study is to determine the feasibility of a uterine sound sparing technique for levonorgestrel 52 mg intrauterine device (IUD) placement. This study will be conducted in three phases. In phase one, the IUD will be placed in standard fashion with a uterine sound to obtain baseline data. Phase two and three are interventional phases that will investigate IUD placement without the use of a uterine sound. In phase two, the IUD will be placed without the use of a uterine sound, but under abdominal ultrasound guidance. In phase three, the IUD will be placed without the use of a uterine sound and without ultrasound guidance. An ultrasound exam will be completed at the end of phase two and three to determine if the IUD was successful placed. To answer the secondary objectives, for all study phases the investigators will measure the procedure time, the participant-reported maximum pain during and 5-minutes post placement and the provider assessment of ease of placement. To determine the exploratory objective of IUD expulsion and perforation rate for a uterine sound sparing IUD placement technique, participants in phases two and three will complete a 30-day phone follow up and 90-day in clinic follow up to evaluate for IUD expulsion or perforation. The investigators hypothesize that the levonorgestrel 52 mg IUD can successfully be inserted without uterine sounding.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Patients undergoing a levonorgestrel 52 mg IUD placement for contraception at a UC Davis outpatient clinic, who have signed consent for placement and are candidates for levonorgestrel 52 mg IUD placement based on the clinical judgement of their UC Davis Ob-Gyn provider.

Exclusion Criteria:

* Women with prior failed IUD placement
* Women with known uterine anomalies or uterine fibroids that distort the uterine cavity
* Women with known cervical stenosis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Successful placement, defined by ultrasound confirmation, of a levonorgestrel 52 mg IUD placement without uterine sounding. | Ultrasound completed at end of IUD placement procedure to determine if successfully placed in the correct location.
  Successful placement without a uterine sound defined as ultrasound confirmation of IUD in the uterine cavity following placement. Outcomes will be compared between experimental phases two and three.

SECONDARY OUTCOMES:
Total time of IUD placement measured in minutes | Measured once on day of IUD placement
  Time measured from the start of the IUD inserter touching the cervix to the removal of the IUD inserter from the cervix in each of the three phases of the study. Outcomes will be compared for each of the three phases.
Participant-reported maximum pain during IUD placement measured with a 100-mm visual analog scale | Measured once on day of IUD placement
  Participants will be handed a 100-mm visual analog scale and asked to mark their pain level. The assessment will be performed immediately following removal of IUD inserter and before the IUD thread is cut. Outcomes will be compared for each of the three phases.
Participant-reported pain 5-minutes post IUD placement, meaured with a 100-mm visual analog scale | Measured once on day of IUD placement
  Participants will be handed a 100-mm visual analog scale and asked to mark their pain level. The assessment will be performed five minutes following removal of the speculum at the end of IUD placement procedure. Outcomes will be compared for each of the three phases.
Provider assessment of ease of placement defined as an easy, moderate or difficult placement. | Measured once on day of IUD placement
  Providers placing the IUD will be asked to rate their assessment of the the ease of the IUD placement procedure as easy, moderate or difficult after completing IUD placement procedure. Outcomes will be compared for each of the three phases.
IUD expulsion and perforation rate during first three months after placement with sound-sparing technique | Measured at time of IUD insertion and three month clinic follow up three months after IUD placement
  An ultrasound exam will be completed on the day of the IUD placement to determine if the IUD is present in the uterine cavity and not perforated outside of the uterine cavity or expelled out of the uterine cavity. Outcomes will be reported for participants in phases two and three.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No